CLINICAL TRIAL: NCT07261020
Title: Comparison of the Effects of Reformer Pilates and Mat Pilates on Certain Physical and Functional Parameters in Women With Lumbar Disc Herniation
Brief Title: The Effectiveness of Pilates in Women With Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar77
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Disc Herniation; Kinesiophobia; Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Kinesiophobia; Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mat exercise group (Experimental): mat pilates exercise
  Interventions: Other: mat pilates
- reformer exercise group (Experimental): reformer pilates exercise
  Interventions: Other: reformer pilates

INTERVENTIONS:
Other: mat pilates — The mat pilates group was given an exercise program consisting of 16 sessions, 2 days a week, for 8 weeks. All exercises were performed as one set of 15 repetitions for the first 2 weeks, 15 repetitions for the 3rd and 4th weeks, and 15 repetitions for the 5th and 6th weeks, with 20 repetitions for the final 2 weeks. Exercise intensity (number of repetitions and level of movement) was gradually increased. Priority was given to core muscles when selecting exercises. The aim was to work the transversus abdominis, multifidus, and gluteus muscles both eccentrically and concentrically, while maintaining spinal stabilization and fostering awareness during movement. The exercise protocol was performed twice a week for 8 weeks, with each session lasting 45 minutes.
  Arms: mat exercise group
Other: reformer pilates — The Reformer Pilates group was assigned an exercise program consisting of 16 sessions, 2 days a week, for 8 weeks. All exercises were performed as one set of 15 repetitions for the first 2 weeks, 15 repetitions for the 3rd and 4th weeks, and 20 repetitions for the 5th and 6th weeks. Exercise intensity (number of repetitions and level of movement) was gradually increased. Priority was given to core muscles when selecting exercises. The aim was to work the transversus abdominis, multifidus, and gluteus muscles both eccentrically and concentrically, while maintaining spinal stabilization and fostering awareness during movement. The exercise protocol consisted of 45-minute sessions, 2 days a week, for 8 weeks.
  Arms: reformer exercise group

SUMMARY:
The aim of the study was to compare the effects of reformer pilates and mat exercise on pain, quality of life and kinesiophobia in female patients with lumbar disc herniation.

DETAILED DESCRIPTION:
The study began with patients diagnosed with lumbar disc herniation. Individuals were invited to participate based on inclusion criteria. Exclusion criteria were used to exclude individuals. Individuals were evaluated twice in this study. Treatment methods were applied. Mat Pilates was applied to one of the diagnosed groups, and reformer Pilates was applied to the other. Twenty participants were assigned to the mat Pilates group and 20 to the equipment Pilates group. A total of 40 patients participated. Pre- and post-treatment assessments were conducted using the Tampa Kinesiophobia Scale, Short Form Quality of Life Scale, and Visual Analog Scale.

ELIGIBILITY:
Inclusion Criteria

* Being between 25 and 60 years of age
* Having been diagnosed with a lumbar disc herniation
* Having agreed to participate in the study

Exclusion Criteria

* Being outside the specified age limits
* Having an orthopedic, neurological, or other condition that prevents exercise

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
quality of life scale short form | 10 weeks
  The scale assessing quality of life consists of 36 questions. It rates health on a scale of 0 to 100, with 0 indicating poor health and 100 indicating good health.
Tampa Kinesiophobia Scale | 10 weeks
  The scale consists of 17 questions. It includes parameters for injury/re-injury and fear-avoidance in work-related activities. Each question is scored using a 4-point Likert scale (1 = strongly disagree, 4 = strongly agree). A total score is calculated by reverse-scoring questions 4, 8, 12, and 16. A higher score is interpreted as indicating a higher level of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça Bilgi, Study Chair — Uskudar University
Locations (1):
- Fone Physio Healthy Living Center, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franks J, Thwaites C, Morris ME. Pilates to Improve Core Muscle Activation in Chronic Low Back Pain: A Systematic Review. Healthcare (Basel). 2023 May 12;11(10):1404. doi: 10.3390/healthcare11101404. PMID 37239690
- [Background] Li Y, Yan L, Hou L, Zhang X, Zhao H, Yan C, Li X, Li Y, Chen X, Ding X. Exercise intervention for patients with chronic low back pain: a systematic review and network meta-analysis. Front Public Health. 2023 Nov 17;11:1155225. doi: 10.3389/fpubh.2023.1155225. eCollection 2023. PMID 38035307
- [Background] Fernandez-Rodriguez R, Alvarez-Bueno C, Cavero-Redondo I, Torres-Costoso A, Pozuelo-Carrascosa DP, Reina-Gutierrez S, Pascual-Morena C, Martinez-Vizcaino V. Best Exercise Options for Reducing Pain and Disability in Adults With Chronic Low Back Pain: Pilates, Strength, Core-Based, and Mind-Body. A Network Meta-analysis. J Orthop Sports Phys Ther. 2022 Aug;52(8):505-521. doi: 10.2519/jospt.2022.10671. Epub 2022 Jun 19. PMID 35722759